CLINICAL TRIAL: NCT05359523
Title: Investigation of the Diagnostic Effect of Ultrasonographic Measurement Values of Upper Back Muscles and Fascia in Patients With Myofascial Pain Syndrome
Brief Title: Ultrasonographic Muscles and Fascia Measurement With Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Assoc.Phd.M.D, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021/10-16
Record Dates: First submitted 2022-04-27; First posted 2022-05-04 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients diagnosed with myofascial pain syndrome (Active Comparator): Ultrasound measurements will be made while the upper back is at rest and during arm movements.
  Interventions: Device: Ultrasonographic measurements of the trapezius and rhomboid muscle and fascia; Other: fascia injection
- Healthy volunteers (Active Comparator): Ultrasound measurements will be made while the upper back is at rest and during arm movements.
  Interventions: Device: Ultrasonographic measurements of the trapezius and rhomboid muscle and fascia

INTERVENTIONS:
Device: Ultrasonographic measurements of the trapezius and rhomboid muscle and fascia — B mode measurements Trapezius and rhomboid muscle thickness and fascial thickness measurement M mode measurements Abduction at 90 and 180 degrees Forward flexion at 90 and 180 degrees
Other: fascia injection — Under ultrasound guidance, a local anesthetic and steroid mixture will be injected into the fascia between the trapezius muscle and the rhomboid muscle.
  Arms: Patients diagnosed with myofascial pain syndrome

SUMMARY:
Pathologies in the trapezius muscle and rhomboid muscle are important in the course and treatment of the disease in patients with myofascial pain syndrome.

DETAILED DESCRIPTION:
In this study, the role of the thickness of these muscles and the shift during movement in the activity and diagnosis of the disease in myofascial pain syndrome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* myofascial pain syndrome

Exclusion Criteria:

* Cervical radiculopathy
* Fibromyalgia
* Shoulder joint disease,
* Peripheral and central nervous system disease
* Polyneuropathy,
* Inflammatory rheumatic disease,
* Malignancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Trapezius muscle and rhomboid muscle thickness | 20 minute
  Trapezius and rhomboid muscle thickness and fascial thickness measurement will be made by ultrasonography at rest.
fascial sliding | 20 minute
  Measurements of the amount of slip measured during the movement of the fascial structures during shoulder and arm movements.
  ultrasonography M-mode measurements Arm from the shoulder joint, cervical lateral flexion, cervical anterior flexion, shoulder elevation

SECONDARY OUTCOMES:
VAS | 6 th month
  visual analog scale (VAS) :for pain. 0: no pain at all, 10: worst pain imaginable
NPDS | 6th month
  Neck and Disability Scale (NPDS):
  The 20-item Neck and Disability Scale is scored on a 10 cm visual analog scale and ranges from 0 to 5 points. The test aims to measure the impact of neck pain on quality of life, functionality, and disability.
SF-12 | 6th month
  Short Form 12 (SF-12): The SF-12 form, which includes scales to assess physical (SF-12-PCS) and mental (SF-12-MCS) status, was created by taking 12 different items from 8 other titles of the SF-36, which is the extended version.
  Interpretation of Scores:
  Utilize the norm-based scoring system to interpret PCS and MCS scores, with a mean of 50 and a standard deviation of 10 in the general population.
  Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Burcu Metin Ökmen, Nilufer, Bursa
  - Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa